CLINICAL TRIAL: NCT01975883
Title: Glycemic Instability of Non-diabetic Patients After Spine Surgery: a Prospective Observational Cohort Study
Brief Title: Glycemic Instability After Spine Surgery
Acronym: GLYRACH
Status: Completed | Type: Observational
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Cyril Dauzac, MD, Beaujon Hospital
Other Study IDs: GLYRACH001
Record Dates: First submitted 2013-10-24; First posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Hyperglycemia
Keywords: Blood Glucose; Postoperative Complications; Spine; Orthopedic surgery
MeSH Terms: conditions — Hyperglycemia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spine surgical patients: Sequential patients scheduled for spine surgery, including degenerative, deformative, tumoral and traumatologic indications are eligible to participate. Exclusion criteria are the following : infection or history of infection of surgical site, past medical history of diabetes mellitus, defined as chronic glucose intolerance either insulin-dependent or non insulin-dependent at the time of operation, and patients with preoperative random BG levels greater than 126 mg/dl considering they could also represent undiagnosed diabetes

SUMMARY:
Analyzing peri operative changes in blood glucose levels from non-diabetic patients undergoing spine surgery

DETAILED DESCRIPTION:
Background: Blood glucose (BG) dysregulation is a well-known situation in medical or surgical severe circumstances. However BG levels following spine surgery have never been described before. Our primary purpose is to measure postoperative changes in BG levels of non-diabetic patients undergoing spine surgery.

Methods: Non-diabetic consecutive adult patients undergoing spine surgery are going to be prospectively included during a 6 months period. BG capillary measures are collected from the preoperative fasting period to the end of postoperative day 3, six times a day. Three main glycemic parameters are calculated: Delta Day 0 (DD0), Day 2 mean (D2), and Hyperglycemic Index (HGI). In the peri operative period, no change in oral intake nor in intravenous fluids is prescribed. Patients are followed-up for three months postoperatively for any early adverse event, requiring or not surgical revision.

ELIGIBILITY:
Inclusion Criteria:

* non diabetic spine surgery candidate

Exclusion Criteria:

* infection or history of infection of surgical site, past medical history of diabetes mellitus, defined as chronic glucose intolerance either insulin-dependent or non insulin-dependent at the time of operation, and patients with preoperative random BG levels greater than 126 mg/dl considering they could also represent undiagnosed diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential patients scheduled for spine surgery in our center, including degenerative, deformative, tumoral and traumatologic indications are eligible to participate.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes in capillary blood glucose levels | 6 times a day, for 3 days after surgery
  Blood glucose levels are measured at the following times: before being lead to the operating room, fasting ; 2 hours after post anesthesia care unit admission ; 30 min before and 2 hours after breakfast, lunch and dinner on the first postoperative day. The same schedule was repeated on the second and the third day after surgery

SECONDARY OUTCOMES:
postoperative local or general, surgical or medical, complication | 6 weeks after surgery for each patient
  Patients are followed on consultation by the medical team six weeks after surgery to determine the occurrence of either surgical revision (due to surgical site infection defined by the criteria of the US Centers for Disease Control and Prevention (CDC), mechanical or neurological complication), or any other early local or general complication such as wound healing impairment, deep venous thromboembolic or cardiovascular event.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Dauzac, MD, Principal Investigator — Hopital Beaujon
Locations (1):
- Hopital Beaujon, Clichy, Hauts-de-Seine, France

REFERENCES:
- [Background] Pili-Floury S, Mitifiot F, Penfornis A, Boichut N, Tripart MH, Christophe JL, Garbuio P, Samain E. Glycaemic dysregulation in nondiabetic patients after major lower limb prosthetic surgery. Diabetes Metab. 2009 Feb;35(1):43-8. doi: 10.1016/j.diabet.2008.06.007. Epub 2008 Nov 26. PMID 19038564
- [Background] Lipshutz AK, Gropper MA. Perioperative glycemic control: an evidence-based review. Anesthesiology. 2009 Feb;110(2):408-21. doi: 10.1097/ALN.0b013e3181948a80. PMID 19194167
- [Background] Pull ter Gunne AF, Cohen DB. Incidence, prevalence, and analysis of risk factors for surgical site infection following adult spinal surgery. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1422-8. doi: 10.1097/BRS.0b013e3181a03013. PMID 19478664